CLINICAL TRIAL: NCT03528668
Title: Patient Receptiveness to Using Virtual Reality as a Distractor From Pain
Brief Title: Patient Receptiveness to Using Virtual Reality
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Paul Arnstein, Clinical Nurse Specialist, Massachusetts General Hospital
Other Study IDs: 2017P002788
Record Dates: First submitted 2018-04-23; First posted 2018-05-18 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Virtual Reality Exposure — Exposure to Virtual Reality program for up to 30 minutes

SUMMARY:
This study will evaluate the acceptability, use, and general effect that exposure to virtual reality has on hospitalized patients reporting at least one discomfort including recent or current moderate-severe pain.

DETAILED DESCRIPTION:
Patients with moderate-severe pain will be approached with approval of nursing staff and front line nurse manager who determine their appropriateness for a trial of virtual reality (VR) exposure for up to 30 minutes. The trial and use of VR will be explained after meeting the inclusion criteria and they will be asked about their level of interest in trying the VR headset. If interested, the subject will indicate their verbal consent to proceed with the VR trial. They will be asked about any baseline discomforts of pain, anxiety/stress or other discomfort; which will be rated on a 0-10 numeric (visual analog) scale. A baseline heart rate will be recorded in beats per minute. The headset will be applied and adjusted for comfort, then the app will be started along with a timer to track the duration of their use up to a maximum of 30 minutes. When the Headset is removed, the duration of use will be noted. The change in post-exposure heart rate (in beats per minute) and discomforts of pain, anxiety/stress or other discomforts (subtracting baseline from 5 minute post-exposure data) will be recorded. Subjects will be asked about the ease of use, whether or not they would use VR again, and for any other comments they would like to express. The headset will be disinfected between patient use.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Inpatients on a general care unit
* Current or recorded moderate to severe pain in past 24 hours

Exclusion Criteria:

* Receiving palliative/end of life care;
* Admitted for treatment of psychiatric or mental health disorder
* History of seizure or stroke
* Legally blind or deaf
* Moderate or severe cognitive impairment
* Head wounds or bandages
* On isolation precautions.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients on adult general care medical/surgical units, regardless of genders will be identified via an existing pain assessment dashboard that allows the investigator to identify patients with 3 or episodes of moderate-severe pain in the prior 24-hour period. The investigator will scan the report for potential subjects in accordance with participating units, inclusion and exclusion criteria. The front-line nurse manager and registered Nurse caring for to patient will be contacted for appropriateness to consider including and the timing when the patient can be approached without interrupting planned tests, treatments or workflow.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain | Change between baseline and 5 minutes after intervention
  Change in subjective report of pain measured on a visual analog scale

SECONDARY OUTCOMES:
Change in Heart Rate | Change between baseline and 5 minutes after intervention
  Change in heart rate measured in beats per minute
Change in Anxiety | Change between baseline and 5 minutes after intervention
  Change in subjective report of anxiety measured on a visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Arnstein, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data will be collected without individual patient identifiers. Patient identifiers will be logged and separately in a locked confidential file.